CLINICAL TRIAL: NCT02755831
Title: Randomized Controlled Trial for a Sleep Study and Targeted CPAP Therapy for Obstructive Sleep Apnea to Reduce the Incidence Adverse Pregnancy Related Outcomes
Brief Title: Targeted CPAP Therapy for Obstructive Sleep Apnea in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, CAPT Dennis Spence, NC, USN, PhD, CRNA, Anesthesia Nurse, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2016.0029
Record Dates: First submitted 2016-03-11; First posted 2016-04-29 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; pregnancy; adverse pregnancy outcomes; continuous positive airway pressure; preeclampsia; gestational diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pre-Eclampsia; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sleep Study + CPAP group (Experimental): Pregnant women in early pregnancy may be randomized to this arm and be assigned Sleep study + CPAP treatment
  Interventions: Device: CPAP
- Standard Prenatal Care group (Other): Pregnant women in early pregnancy may be randomized to this arm and will receive standard prenatal care without CPAP treatment.
  Interventions: Other: Pre-natal care

INTERVENTIONS:
Device: CPAP — Continuous Positive Airway Pressure (CPAP) Therapy for Obstructive Sleep Apnea
  Arms: Sleep Study + CPAP group
Other: Pre-natal care — Standard Pre-Natal Care
  Arms: Standard Prenatal Care group

SUMMARY:
Prospective, randomized controlled trial. Pregnant women in early pregnancy will be randomized to either the Sleep Study + CPAP (Continuous Positive Airway Pressure Therapy) group or to a Standard Prenatal Care group. Subjects in the Sleep Study + CPAP group will complete a sleep study (WatchPAT-200, Itamar Medical, Inc.) and have CPAP initiated if the Apnea Hypopnea Index (AHI) ≥5 as indicated, in early and late pregnancy, whereas the other group will receive standard prenatal care. All subjects will complete a sleep study again between 8 to 12 weeks postpartum.

DETAILED DESCRIPTION:
Objective/Hypothesis: The purpose of this study is to determine if parturients identified as high risk for obstructive sleep apnea (OSA; defined as an apnea hypopnea index [AHI] ≥5 events/hour) who are randomized to receive an unattended sleep study during early and late pregnancy (early = between 6 and 16 weeks; late = between 27 and 33 weeks) plus initiation of CPAP therapy if the AHI ≥5 events/hour and standard prenatal care have a decreased incidence of adverse pregnancy outcomes (defined as a composite variable which includes gestational hypertension, preeclampsia, eclampsia, gestational diabetes, preterm birth, low birth weight, or stillbirth) at the time of delivery when compared to a group who receives standard prenatal care only (no sleep study and CPAP initiation). At 8 to 12 months postpartum subjects in both groups will complete a sleep study.

ELIGIBILITY:
Inclusion Criteria

1. At least one of the following risk factors for OSA: prepregnancy BMI ≥ 30kg/m2, chronic hypertension, pregestational diabetes, twin gestation, or a history of prior pregnancy affected by: preeclampsia, eclampsia or fetal growth restriction.
2. Between 6 and 16 weeks gestation at time of enrollment.

Exclusion Criteria

1. Current diagnosis and treatment of OSA.
2. Patient refusal to randomization.
3. Permanent Pacemaker (interfere with WATCHPAT sleep study).
4. Currently taking alpha blockers or nitrates (interfere with WATCHPAT sleep study).
5. Coronary artery disease or congestive heart failure or cardiomyopathy.
6. Not delivering and completing their postpartum visit at Naval Medical Center San Diego (NMCSD).
7. Inability to read or understand the consent.
8. <18 years of age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Spence, PhD, Study Director — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to submit manuscripts to appropriate journals and present data at appropriate conferences

REFERENCES:
- [Background] Poyares D, Guilleminault C, Hachul H, Fujita L, Takaoka S, Tufik S, Sass N. Pre-eclampsia and nasal CPAP: part 2. Hypertension during pregnancy, chronic snoring, and early nasal CPAP intervention. Sleep Med. 2007 Dec;9(1):15-21. doi: 10.1016/j.sleep.2007.04.019. Epub 2007 Jul 20. PMID 17644475
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Young T, Finn L, Peppard PE, Szklo-Coxe M, Austin D, Nieto FJ, Stubbs R, Hla KM. Sleep disordered breathing and mortality: eighteen-year follow-up of the Wisconsin sleep cohort. Sleep. 2008 Aug;31(8):1071-8. PMID 18714778
- [Background] Young T, Palta M, Dempsey J, Peppard PE, Nieto FJ, Hla KM. Burden of sleep apnea: rationale, design, and major findings of the Wisconsin Sleep Cohort study. WMJ. 2009 Aug;108(5):246-9. PMID 19743755
- [Background] Memtsoudis SG, Sun X, Chiu YL, Nurok M, Stundner O, Pastores SM, Mazumdar M. Utilization of critical care services among patients undergoing total hip and knee arthroplasty: epidemiology and risk factors. Anesthesiology. 2012 Jul;117(1):107-16. doi: 10.1097/ALN.0b013e31825afd36. PMID 22634871
- [Background] Luque-Fernandez MA, Bain PA, Gelaye B, Redline S, Williams MA. Sleep-disordered breathing and gestational diabetes mellitus: a meta-analysis of 9,795 participants enrolled in epidemiological observational studies. Diabetes Care. 2013 Oct;36(10):3353-60. doi: 10.2337/dc13-0778. PMID 24065843
- [Background] Ding XX, Wu YL, Xu SJ, Zhang SF, Jia XM, Zhu RP, Hao JH, Tao FB. A systematic review and quantitative assessment of sleep-disordered breathing during pregnancy and perinatal outcomes. Sleep Breath. 2014 Dec;18(4):703-13. doi: 10.1007/s11325-014-0946-4. Epub 2014 Feb 12. PMID 24519711
- [Background] Pamidi S, Pinto LM, Marc I, Benedetti A, Schwartzman K, Kimoff RJ. Maternal sleep-disordered breathing and adverse pregnancy outcomes: a systematic review and metaanalysis. Am J Obstet Gynecol. 2014 Jan;210(1):52.e1-52.e14. doi: 10.1016/j.ajog.2013.07.033. Epub 2013 Aug 2. PMID 23911687
- [Background] Louis J, Auckley D, Miladinovic B, Shepherd A, Mencin P, Kumar D, Mercer B, Redline S. Perinatal outcomes associated with obstructive sleep apnea in obese pregnant women. Obstet Gynecol. 2012 Nov;120(5):1085-92. doi: 10.1097/AOG.0b013e31826eb9d8. PMID 23090526
- [Background] American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: an updated report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2014 Feb;120(2):268-86. doi: 10.1097/ALN.0000000000000053. No abstract available. PMID 24346178
- [Background] Ankichetty SP, Angle P, Joselyn AS, Chinnappa V, Halpern S. Anesthetic considerations of parturients with obesity and obstructive sleep apnea. J Anaesthesiol Clin Pharmacol. 2012 Oct;28(4):436-43. doi: 10.4103/0970-9185.101895. PMID 23225920
- [Background] Reutrakul S, Zaidi N, Wroblewski K, Kay HH, Ismail M, Ehrmann DA, Van Cauter E. Interactions between pregnancy, obstructive sleep apnea, and gestational diabetes mellitus. J Clin Endocrinol Metab. 2013 Oct;98(10):4195-202. doi: 10.1210/jc.2013-2348. Epub 2013 Aug 21. PMID 23966237
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Louis JM, Mogos MF, Salemi JL, Redline S, Salihu HM. Obstructive sleep apnea and severe maternal-infant morbidity/mortality in the United States, 1998-2009. Sleep. 2014 May 1;37(5):843-9. doi: 10.5665/sleep.3644. PMID 24790262
- [Background] Facco FL, Ouyang DW, Zee PC, Grobman WA. Sleep disordered breathing in a high-risk cohort prevalence and severity across pregnancy. Am J Perinatol. 2014 Nov;31(10):899-904. doi: 10.1055/s-0033-1363768. Epub 2014 Feb 10. PMID 24515622
- [Background] Pien GW, Pack AI, Jackson N, Maislin G, Macones GA, Schwab RJ. Risk factors for sleep-disordered breathing in pregnancy. Thorax. 2014 Apr;69(4):371-7. doi: 10.1136/thoraxjnl-2012-202718. Epub 2013 Nov 21. PMID 24262432
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Morgenthaler TI, Aurora RN, Brown T, Zak R, Alessi C, Boehlecke B, Chesson AL Jr, Friedman L, Kapur V, Maganti R, Owens J, Pancer J, Swick TJ; Standards of Practice Committee of the AASM; American Academy of Sleep Medicine. Practice parameters for the use of autotitrating continuous positive airway pressure devices for titrating pressures and treating adult patients with obstructive sleep apnea syndrome: an update for 2007. An American Academy of Sleep Medicine report. Sleep. 2008 Jan;31(1):141-7. doi: 10.1093/sleep/31.1.141. PMID 18220088
- [Background] Guilleminault C, Palombini L, Poyares D, Takaoka S, Huynh NT, El-Sayed Y. Pre-eclampsia and nasal CPAP: part 1. Early intervention with nasal CPAP in pregnant women with risk-factors for pre-eclampsia: preliminary findings. Sleep Med. 2007 Dec;9(1):9-14. doi: 10.1016/j.sleep.2007.04.020. Epub 2007 Jul 17. PMID 17644420
- [Background] Whitehead C, Tong S, Wilson D, Howard M, Walker SP. Treatment of early-onset preeclampsia with continuous positive airway pressure. Obstet Gynecol. 2015 May;125(5):1106-1109. doi: 10.1097/AOG.0000000000000508. PMID 25774926
- [Background] Facco F. Sleep-disordered breathing in pregnancy: a brief summary of current knowledge. BJOG. 2014 Dec;121(13):1694. doi: 10.1111/1471-0528.12888. Epub 2014 May 30. No abstract available. PMID 24889020
- [Background] Izci-Balserak B, Pien GW. Sleep-disordered breathing and pregnancy: potential mechanisms and evidence for maternal and fetal morbidity. Curr Opin Pulm Med. 2010 Nov;16(6):574-82. doi: 10.1097/MCP.0b013e32833f0d55. PMID 20859210
- [Background] Volna J, Kemlink D, Kalousova M, Vavrova J, Majerova V, Mestek O, Svarcova J, Sonka K, Zima T. Biochemical oxidative stress-related markers in patients with obstructive sleep apnea. Med Sci Monit. 2011 Sep;17(9):CR491-7. doi: 10.12659/msm.881935. PMID 21873945
- [Background] Lyall F, Robson SC, Bulmer JN. Spiral artery remodeling and trophoblast invasion in preeclampsia and fetal growth restriction: relationship to clinical outcome. Hypertension. 2013 Dec;62(6):1046-54. doi: 10.1161/HYPERTENSIONAHA.113.01892. Epub 2013 Sep 23. PMID 24060885
- [Background] Fung AM, Wilson DL, Lappas M, Howard M, Barnes M, O'Donoghue F, Tong S, Esdale H, Fleming G, Walker SP. Effects of maternal obstructive sleep apnoea on fetal growth: a prospective cohort study. PLoS One. 2013 Jul 24;8(7):e68057. doi: 10.1371/journal.pone.0068057. Print 2013. PMID 23894293
- [Background] Young T, Evans L, Finn L, Palta M. Estimation of the clinically diagnosed proportion of sleep apnea syndrome in middle-aged men and women. Sleep. 1997 Sep;20(9):705-6. doi: 10.1093/sleep/20.9.705. PMID 9406321
- [Background] Reid J, Glew RA, Skomro R, Fenton M, Cotton D, Olatunbosun F, Gjevre J, Guilleminault C. Sleep disordered breathing and gestational hypertension: postpartum follow-up study. Sleep. 2013 May 1;36(5):717-721B. doi: 10.5665/sleep.2634. PMID 23633754
- [Background] Hermes W, Tamsma JT, Grootendorst DC, Franx A, van der Post J, van Pampus MG, Bloemenkamp KW, Porath M, Mol BW, de Groot CJ. Cardiovascular risk estimation in women with a history of hypertensive pregnancy disorders at term: a longitudinal follow-up study. BMC Pregnancy Childbirth. 2013 Jun 4;13:126. doi: 10.1186/1471-2393-13-126. PMID 23734952
- [Background] Chen YH, Kang JH, Lin CC, Wang IT, Keller JJ, Lin HC. Obstructive sleep apnea and the risk of adverse pregnancy outcomes. Am J Obstet Gynecol. 2012 Feb;206(2):136.e1-5. doi: 10.1016/j.ajog.2011.09.006. Epub 2011 Sep 16. PMID 22000892
- [Background] Facco FL, Ouyang DW, Zee PC, Grobman WA. Development of a pregnancy-specific screening tool for sleep apnea. J Clin Sleep Med. 2012 Aug 15;8(4):389-94. doi: 10.5664/jcsm.2030. PMID 22893769
- [Background] Hedner J, Pillar G, Pittman SD, Zou D, Grote L, White DP. A novel adaptive wrist actigraphy algorithm for sleep-wake assessment in sleep apnea patients. Sleep. 2004 Dec 15;27(8):1560-6. doi: 10.1093/sleep/27.8.1560. PMID 15683148
- [Background] Penzel T, Kesper K, Pinnow I, Becker HF, Vogelmeier C. Peripheral arterial tonometry, oximetry and actigraphy for ambulatory recording of sleep apnea. Physiol Meas. 2004 Aug;25(4):1025-36. doi: 10.1088/0967-3334/25/4/019. PMID 15382839
- [Background] Ahmadi N, Chung SA, Gibbs A, Shapiro CM. The Berlin questionnaire for sleep apnea in a sleep clinic population: relationship to polysomnographic measurement of respiratory disturbance. Sleep Breath. 2008 Mar;12(1):39-45. doi: 10.1007/s11325-007-0125-y. PMID 17684781
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Rogers AE, Caruso CC, Aldrich MS. Reliability of sleep diaries for assessment of sleep/wake patterns. Nurs Res. 1993 Nov-Dec;42(6):368-72. PMID 8247821
- [Background] Haythornthwaite JA, Hegel MT, Kerns RD. Development of a sleep diary for chronic pain patients. J Pain Symptom Manage. 1991 Feb;6(2):65-72. doi: 10.1016/0885-3924(91)90520-e. PMID 2007794
- [Background] Finkel KJ, Searleman AC, Tymkew H, Tanaka CY, Saager L, Safer-Zadeh E, Bottros M, Selvidge JA, Jacobsohn E, Pulley D, Duntley S, Becker C, Avidan MS. Prevalence of undiagnosed obstructive sleep apnea among adult surgical patients in an academic medical center. Sleep Med. 2009 Aug;10(7):753-8. doi: 10.1016/j.sleep.2008.08.007. Epub 2009 Jan 30. PMID 19186102
- [Derived] Kalkhoff SM, Lutgendorf MA, Morrison TC, Han T, Spence DL. A randomized controlled trial of sleep study surveillance with targeted autoregulated positive airway pressure therapy for obstructive sleep apnea in pregnancy. Am J Obstet Gynecol MFM. 2022 May;4(3):100571. doi: 10.1016/j.ajogmf.2022.100571. Epub 2022 Jan 17. PMID 35051670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment. There were 714 women assessed for eligibility with N = 193 enrolled; n = 100 allocated to treatment group and n = 93 to the control group. In the treatment group there were n = 3 and n = 3 in the control group, respectively, loss to follow-up. The final analysis included n = 97 in the treatment group and n = 90 in the control group.
Period: Overall Study
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group
Started | 100 | 93
Completed | 97 | 90
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group | Total
Number analyzed (Participants) | 100 | 93 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 93 | 193
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.8) | 28.8 (5.2) | 29 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 93 | 193
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 16 | 37
  White | 43 | 46 | 89
  More than one race | 20 | 16 | 36
  Unknown or Not Reported | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 100 | 93 | 193
Pre-Pregnancy BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.5 (7) | 33.3 (6.8) | 33.9 (7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Pregnancy Outcomes
Description: Number of participants with adverse pregnancy outcomes (composite outcome includes: gestational hypertension, preeclampsia, eclampsia, gestational diabetes, preterm delivery, low birth weight, or stillbirth)
Time Frame: time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group
Number analyzed (Participants) | 97 | 90
Participants | 45 | 39
Statistical Analysis 1: Comparison: Sleep Study + CPAP Group vs Standard Prenatal Care Group; Fisher's Exact Test; Test type: Superiority; p < 0.05, Fisher Exact

2. Secondary Outcome: Incidence of Obstructive Sleep Apnea (OSA) in Early Pregnancy - Treatment Group Only (6-16 Weeks)
Description: Incidence of OSA severity in early pregnancy (6-16 weeks) in treatment group only. Data were not collected for Control group at this time point.
Time Frame: early pregnancy (6-16 weeks)
Population: Friedman's test was used to analyze differences in sleep study results at the three time points in experimental group. If significant differences are found in sleep study results a post hoc Wilcoxon Ranked Sign test will be used to compare differences at individual time points. Data were not collected for Control group at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Study + CPAP Group
Number analyzed (Participants) | 93
Participants
  No OSA | 89
  mild OSA | 3
  moderate OSA | 0
  severe OSA | 1
Statistical Analysis 1: Comparison: Sleep Study + CPAP Group; Test type: Other; p < .05, Friedman test; Friedman's test was used to analyze differences with a post hoc Wilcoxon Ranked Sign test to compare differences at individual time points

3. Secondary Outcome: Incidence of OSA in Late Pregnancy- Treatment Group Only (27-33 Weeks)
Description: Incidence and severity of OSA in late pregnancy- treatment group only (27-33 weeks). Data were not collected for Control group at this time point
Time Frame: 27-33 weeks
Population: Incidence and Severity of OSA in Late Pregnancy. Outcome data was only collected in the treatment group. Data were not collected for Control group at this time point
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Study + CPAP Group
Number analyzed (Participants) | 92
Participants
  No OSA | 81
  Mild OSA | 11
  Moderate OSA | 0
  Severe OSA | 0
Statistical Analysis 1: Comparison: Sleep Study + CPAP Group; Test type: Other; p < 0.05, Friedman; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Incidence of OSA at 8 to 12 Weeks Postpartum in Treatment and Control Group
Description: Incidence and severity of OSA at 8 to 12 weeks postpartum in treatment and control group.
Time Frame: 8-12 weeks postpartum
Population: Incidence and Severity of OSA at 8-12 weeks postpartum. This is the only time point in which both groups completed sleep studies.
Measure: Count of Participants; unit: Participants
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group
Number analyzed (Participants) | 89 | 80
Participants
  No OSA | 72 | 69
  mild OSA | 14 | 9
  Moderate OSA | 2 | 2
  Severe OSA | 1 | 0
Statistical Analysis 1: Comparison: Sleep Study + CPAP Group vs Standard Prenatal Care Group; Test type: Other; p < 0.05, Friedman Test; Friedman's test was used to analyze differences with a post hoc Wilcoxon Ranked Sign test to compare differences in treatment group only

5. Secondary Outcome: Hospital Costs at Time of Delivery
Description: Hospital costs at time of delivery in treatment and control group.
Time Frame: Hospital costs at time of delivery
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group
Number analyzed (Participants) | 97 | 90
dollars | 12185 [11155 to 13215] | 12607 [11210 to 14004]
Statistical Analysis 1: Comparison: Sleep Study + CPAP Group vs Standard Prenatal Care Group; Test type: Superiority; p < 0.05, t-test, 2 sided; T-test used to compare mean difference in hospital costs at time of delivery

ADVERSE EVENTS:
Time Frame: Adverse data collected after time of enrollment to study completion ( February 20, 2017 - October 14, 2019). Subjects were enrolled starting at 6 to 12 weeks gestation and were followed until approximately 3 months postpartum (8 to 12 weeks postpartum).
Description: No adverse events occurred
Arm/Group | Sleep Study + CPAP Group | Standard Prenatal Care Group
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/90
Other Adverse Events (participants affected / at risk) | 0/97 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT02755831/Prot_SAP_000.pdf